CLINICAL TRIAL: NCT06204939
Title: Extended Pouch Gastric Bypass vs One-anastomosis Gastric Bypass in Patients With a BMI of 45 or Higher: a Randomized Controlled Trial
Brief Title: Extended Pouch Gastric Bypass vs One-anastomosis Gastric Bypass in Patients With BMI≥45
Acronym: EXPANT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: L. van Hogezand (Other)
Collaborators: Rijnstate Hospital (Other)
Responsible Party: Sponsor-Investigator, L. van Hogezand, Coordinating investigator, St. Antonius Hospital
Organization: St. Antonius Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2023-12-08; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Bariatric Surgery Candidate
Keywords: bariatric; gastric bypass; extended pouch; one anastomosis

STUDY DESIGN:
Intervention Model Description: Single blinded randomized controlled trial
Who Masked: Participant
Masking Description: Patients will be randomized single blinded for one of two study arms/procedures. 3 years post-operative unblinding will be done for participants wishing this.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extended Pouch gastric bypass (EPGB) (Other): Classic gastric bypass with 2 anastomoses but with an extended pouch of 12-15cm and a biliary limb of 150cm.
  Interventions: Procedure: Randomizing for EPGB procedure
- One Anastomosis gastric bypass (OAGB) (Other): Gastric bypass with 1 anastomosis and an extended pouch of 12-15cm and a biliary limb of 150cm.
  Interventions: Procedure: Randomizing for OAGB procedure

INTERVENTIONS:
Procedure: Randomizing for EPGB procedure — Classic gastric bypass with 2 anastomoses but with an extended pouch of 12-15cm and a biliary limb of 150cm.
  Patients will be single blinded randomized for one of the two procedures. 125 patients will undergo EPGB and 125 patients will undergo OAGB.
  Pre-operatively, 6 months post-op and yearly post-op we will collect: weight, complications, revisions, comorbidities, blood samples and questionnaires.
  Arms: Extended Pouch gastric bypass (EPGB)
Procedure: Randomizing for OAGB procedure — Gastric bypass with 1 anastomosis and an extended pouch of 12-15cm and a biliary limb of 150cm.
  Patients will be single blinded randomized for one of the two procedures. 125 patients will undergo EPGB and 125 patients will undergo OAGB.
  Pre-operatively, 6 months post-op and yearly post-op we will collect: weight, complications, revisions, comorbidities, blood samples and questionnaires.
  Arms: One Anastomosis gastric bypass (OAGB)

SUMMARY:
The classic RYGB is in most patients with a BMI ≥45 technically not feasible. Two alternatives are the Extended Pouch Gastric Bypass and the One Anastomosis gastric bypass. In this single blinded randomized controlled trial the investigators aim to establish which technique leads to more weightloss in bariatric patients with a BMI ≥45.

DETAILED DESCRIPTION:
Obesity is of increasing incidence worldwide. With it come major social-economical, medical and psychological problems which lead to high healthcare costs. Bariatric surgery is the most efficient treatment for morbid obesity, with the Roux-en-Y gastric bypass (RYGB) and sleeve gastrectomy (GS) being the most performed.

The RYGB is preferable since this technique seems to lead to more reduction of obesity related comorbidities (DM2) and more weightloss in the long term. However, the RYGB is technically less feasible in patients with a BMI ≥45, due to less intra-abdominal space (excess fat in mesenterium) to connect the anastomosis tension-free.

An alternative for the RYGB are the Extended Pouch gastric bypass (EPGB) and the One-Anastomosis gastric bypass (OAGB). These techniques both involve an extended pouch which makes it easier to connect the anastomosis tension-free.

Furthermore, the extended pouch in the EPGB and OAGB could provide slower passage of food and stretches less on the longer term than the 'normal size'pouch in the RYGB, possibly leading to more weightloss (1,2).

Previous studies comparing the EPGB and RYGB showed more weightloss in patient undergoing EPGB and less weight gain in the long term (3). Other studies comparing the OAGB, RYGB and GS showed non-inferiority or even superiority of the OAGB for weightloss and remission of obesity related comorbidities as diabetes mellitus type 2 (DM2) and obstructive sleep apnea syndrome (OSAS) (4,5,6,7).

Theoretically the OAGB is a simpler procedure which reduces the risk of internal herniation and anastomotic leakage, since only one anastomosis is made (6,8) Only performing one anastomosis leads to less operating time, shorter time of anesthesia, and less usage of staple material. Which possibly makes this a safer and cheaper procedure.

Both techniques, EPGB and OAGB, seem to be adequate alternatives for the RYGB in patients with a BMI of 45 or higher. As of yet, the two techniques haven't been compared one to one. In this single blinded randomized controlled trial the investigators aim to establish which technique leads to more weightloss in bariatric patients with a BMI ≥45.

ELIGIBILITY:
Inclusion criteria:

* BMI≥45
* Bariatric guidelines Fried
* Age 18-65
* Dedication to guided preoperative program
* Intention to follow full postoperative program

Exclusion criteria:

* Secondary bariatric procedure
* Medical(-related) cause for morbid obesity or fast weight gain (e.g. Cushing or medication related)
* Inflammatory Bowel Disease (M. Crohn or Colitis Ulcerosa)
* Renal function disorder (MDRD <30) or liver disease
* Anticipated absence of yearly medical follow up
* Does not speak Dutch language
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Weightloss short term | 1, 3 and 5 years postoperatively
  percentage excess weight loss

SECONDARY OUTCOMES:
Weightloss long term | 5-10 years postoperatively
  percentage excess weight loss
Complications short term | up to 30 days postoperatively
  bleeding, leakage, infections, intra-abdominal abcess, readmission, mortality
Complications long term | from 30 days until 10 years postoperatively
  vitamin/electrolyte deficiencies, internal herniation, marginal ulceration
Revision of the bypass | until 10 years postoperatively
  Surgical revision of bypass
Comorbidities | until 10 years postoperatively
  Reduction of obesity-related comorbidites: diabetes mellitus type 2, hypertension, hypercholesterolemia, joint aches en obstructive sleep apnea syndrome
Deficiencies in blood - red blood count | until 10 years postoperatively
  Blood samples: red blood count
Deficiencies in blood - vitamins | until 10 years postoperatively
  Blood samples vitamins
Deficiencies in blood - electrolytes | until 10 years postoperatively
  Blood samples: electrolytes
Reflux/dumping questionnaire | until 10 years postoperatively
  Questionnaires for reflux and dumping complaints. scales 0-10, higher is worse outcome
Health related quality of life questionnaire | until 10 years postoperatively
  Questionnaires on HrQoL and patient satisfaction of procedure, scales 0-5 and 0-10, higher is worse outcome
Peroperative complications | until 10 years postoperatively
  Peroperative complications: bleeding, iatrogenic complications
Number of patients with peroperative conversion to sleeve | until 10 years postoperatively
  Conversion to sleeve when bypass not feasible

CONTACTS AND LOCATIONS:
Overall Officials: Wouter Derksen, MD PhD, Principal Investigator — St. Antonius Hospital

IPD SHARING:
Plan to Share IPD: No
No sharing.